CLINICAL TRIAL: NCT04070521
Title: Observational Study of EEG Monitoring of Patients in the Emergency Department
Brief Title: EEG Monitoring in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Patrick L. Purdon, Nathaniel M. Sims Endowed Chair in Anesthesia Innovation and Bioengineering, Massachusetts General Hospital
Other Study IDs: 2018P002483
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Drug Overdose; Substance Abuse; Alcohol Abuse
Keywords: Electroencephalogram; Opioids; Alcohol; Benzodiazepines; Alpha-2 agonists; Propofol; Ketamine; Marijuana; Neuromechanisms of intoxicants
MeSH Terms: conditions — Drug Overdose; Substance-Related Disorders; Alcoholism; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational EEG Monitoring
  Interventions: Other: Observational EEG Monitoring

INTERVENTIONS:
Other: Observational EEG Monitoring — Subjects will be monitored with electroencephalogram (EEG) after arriving to the Emergency Department with suspected overdose

SUMMARY:
This study seeks to investigate whether drug effects in suspected overdose patients could be identified using the electroencephalogram (EEG). From previous work it is known that different classes of anesthetic drugs have specific "EEG signatures" related to the drug mechanisms. Many of the drugs of abuse that are frequently encountered in overdose patients are similar or identical to anesthetic drugs. The hypothesis for this study is that the EEG could be used to characterize the brain effects of intoxicants using EEG in the ED setting. Such monitoring could one day help clinicians and first responders at the point-of-care make more informed decisions to improve the care of overdose patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older who present to the ED with suspected use of a potential drug of abuse

Exclusion Criteria:

* Hemodynamic instability or other acute medical condition for which the primary treating team does not thing it would be appropriate or safe for the study staff to approach the patient
* The patient has an overt head trauma or deformity of the face which would preclude application of the forehead EEG monitoring lead
* The patient has dermatological issues or skin conditions on the forehead
* The patient has known dementia and/or mental impairment
* The patient is a prisoner
* The patient is an employee or student at one of the study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older who present to the ED with suspected use of a potential drug of abuse.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) | 24 hours
  Subject EEG activity following arrival to Emergency Department with suspected overdose, including EEG waveform, spectrum, spectrogram, and power in the slow (0.1-1 Hz), delta (1 to 4 Hz), theta (4 to 8 Hz), alpha (8 to 12 Hz), beta (12 to 25 Hz), and gamma (25 to 70 Hz) bands.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick L Purdon, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.